CLINICAL TRIAL: NCT02134470
Title: Diagnostic Relevance of Salivary Testosterone Concentrations After Exogene Low-dose Hormone Application as a Screening Method for in Doping Control.
Brief Title: Diagnostic Relevance of Salivary Testosterone Concentrations in Doping Control.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paracelsus Medical University (Other)
Collaborators: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Martin Schoenfelder, Head of Institute, Research Institute of Molecular Sports Medicine and Rehabilitation, Paracelsus Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BISP-SALIVA-2014
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Circadian; Exercise; Testosterone
Keywords: saliva; blood; urine
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone (Experimental): Chemical testing of saliva is an objective method to quantify steroid hormones. Recent studies indicate that salivary testosterone is significantly higher than in other body fluids. Therefore, saliva may serve as pre-screening parameter to select suspicious cases for further target evaluation. The aim of the present project is to detect administered testosterone in saliva and compare these levels to those in blood and urine. Therefore, each participant represents its own control.
  Interventions: Drug: Testosterone supplementation

INTERVENTIONS:
Drug: Testosterone supplementation — Low-dose testosterone supplementation will be facilitated by using hormone patches. For pharmacokinetic aspects circadian profiles of saliva/blood/urine will be measured under native conditions and under exogene hormone application. In addition, cross-reactivity of a standardized exercise bout and hormone application will be of further interest.

SUMMARY:
It is generally accepted that chemical testing of biologic fluids is the most objective means of diagnosis of drug use. In recent years saliva has attracted much attention. The prime advantage of saliva is that it offers non-invasive, stress-free and real-time repeated sampling whereas blood collection is undesirable, difficult and expensive. In addition, it is known that androgens such as testosterone can be assayed in saliva, as these steroids pass the endothelial-epithelial barriers by passive diffusion. Nevertheless, the correlations of blood, urine and saliva concentrations are not well documented. In recent reviews, it is pointed out that salivary hormone analysis could be a promising method for sports medicine and doping control, but much work is needed before the use of saliva samples in this area receives the acceptance. According to recent studies the increase of testosterone concentration in saliva is significantly higher than alterations of steroid concentrations (or ratios) in blood or urine. Saliva concentration may therefore serve as screening parameter to select suspicious cases for further target evaluation (e.g. by IRMS). This may be beneficial to identify cases of transdermal administration of low steroid doses. It is therefore the aim of the present project to detect administered testosterone in saliva and compare these levels to those in blood and urine. The intention is not to detect high dosage but low dosage abuse of testosterone, as a single-dose by patch application. From the practical point of view saliva could offer a complementary specimen for a pre-screening of testosterone. So it could be assumed that salivary testosterone exceed upon plasma and/or urine levels. So the present study could be the base for a new method to preselect the suspicious samples for testosterone abuse.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* informed consent

Exclusion Criteria:

* any metabolic, cardiovascular, pulmonary disorder
* neoplastic or hormonal disorders
* active sports competitor
* disorders which hinder cycling ergometry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Salivary testosterone concentration | 2 weeks
  Salivary testosterone concentration will be quantified in relation to circadian time, exercise, and external low-dose hormone application.

SECONDARY OUTCOMES:
Serum testosterone | 2 weeks
  Serum testosterone concentration (free/bound) will be quantified in relation to circadian time, exercise, and external low-dose hormone application.
Circulating microRNA in blood plasma | 2 weeks
  Circulating microRNA in blood plasma will be screened in relation to circadian time, exercise, and external low-dose hormone application.

OTHER OUTCOMES:
Testosterone in hairs | 4 weeks
  At onset, 2 weeks and 4 weeks after testosterone application steroid hormone concentration will be quantified in scalp hair.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schönfelder, Dr., Principal Investigator — Paracelsus Medical Private University Salzburg, AUT; Hande Hofmann, Dr., Principal Investigator — Technische Universität München, GER; Detlef Thieme, Dr., Principal Investigator — Institute of Doping Analysis und Sports Biochemistry Dresden in Kreischa, GER
Locations (1):
- Technische Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Background] Schonfelder M, Hofmann H, Anielski P, Thieme D, Oberhoffer R, Michna H. Gene expression profiling in human whole blood samples after controlled testosterone application and exercise. Drug Test Anal. 2011 Oct;3(10):652-60. doi: 10.1002/dta.360. PMID 22031502
- [Background] Thieme D, Rautenberg C, Grosse J, Schoenfelder M. Significant increase of salivary testosterone levels after single therapeutic transdermal administration of testosterone: suitability as a potential screening parameter in doping control. Drug Test Anal. 2013 Nov-Dec;5(11-12):819-25. doi: 10.1002/dta.1536. Epub 2013 Oct 25. PMID 24167110
- See also: Institute of Preventive Pediatrics — http://www.praeventive-paediatrie.sg.tum.de/forschung/